CLINICAL TRIAL: NCT01698203
Title: Postoperative Analgesia After Thoracotomy Without Thoracic Epidural Analgesia: Continuous Wound Catheter Analgesia Associated With Intravenous Morphine Patient-Controlled-Analgesia (PCA)
Brief Title: Continuous Wound Catheter Analgesia Associated With Intravenous Morphine PCA After Thoracotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 5277
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Pain; Thoracotomy
MeSH Terms: conditions — Pain | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ropivacaine (Experimental)
  Interventions: Drug: ropivacaine 0.75% - device : wound catheter Silver™ 19 cm and Easypump™ 400 mL (BBraun); Drug: ropivacaine 0.2% - device : wound catheter Silver™ 19 cm and Easypump™ 400 mL (BBraun)
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ropivacaine 0.75% - device : wound catheter Silver™ 19 cm and Easypump™ 400 mL (BBraun) — The group ropivacaine, an initial bolus of 0.75% ropivacaine at a volume of 0.1 ml / kg is first administered to the patient directly on the catheter.
  Arms: ropivacaine
Drug: Placebo — In the placebo group, an initial bolus of saline 9 ‰ to a volume of 0.1 ml / kg will first be administered to the patient directly to the catheter. The patient will then continuous administration of saline 9 ‰ during the first 48 postoperative hours, using a diffuser extensible elastomeric ™ Easypump a volume of 400 mL to 460 mL filled of this solution, a flow rate of 9.53 ml / hour.
  Arms: placebo
Drug: ropivacaine 0.2% - device : wound catheter Silver™ 19 cm and Easypump™ 400 mL (BBraun) — The patient will then ongoing administration of ropivacaine 0.2% during the first 48 postoperative hours, using a diffuser extensible elastomeric ™ Easypump a volume of 400 mL to 460 mL filled (B Braun) of this solution, a flow rate of 9.53 ml / hour
  Arms: ropivacaine

SUMMARY:
Objective: Epidural analgesia is the gold standard for post-thoracotomy pain relief but is contraindicated in certain patients. An alternative is continuous wound catheter analgesia. We will investigate whether ropivacaine, administered through a wound catheter placed by the surgeon, will reduce postoperative pain. Methods: In a randomized double-blind study, adult patients with a wound catheter placed by the thoracic surgeon after thoracotomy will be randomly assigned to receive through this catheter, either a 0.1 mL/kg bolus of 0.75% ropivacaine, followed by a continuous infusion of 0.2% ropivacaine at 10 mL/h for 48 h, or saline at the same scheme of administration. Patients will also benefit from patient-controlled analgesia with intravenous morphine (bolus 1 mg, lockout time 7 min), paracetamol, and nefopam. The primary endpoint will be total morphine consumption. Secondary endpoints will be pain intensity on a visual analog scale at rest and on coughing and side effects during the first 48 postoperative hours. Surgeons, anesthesiologists, and all the nurses and caring staff involved in this study will be blinded. Solutions of saline and ropivacaine will be prepared identically by the central pharmacy, without any possible identification of the product.

ELIGIBILITY:
Inclusion Criteria:

Patients scheduled for thoracotomy who presented with contraindications to TEA.

Contraindications to TEA are :

* Patient's refusal after informations about advantages and risks of the technique
* Anti platelets treatment that can't be discontinued
* Anticoagulants at a curative dosage
* haemostasis and/or coagulation disorders: thrombopenia < 100.000/mm3, ACT > 1,5 / control, PTT < 75%
* Systemic or local infection of the puncture point
* 2 and 3 grade atrio-ventricular heart block without pacing
* Severe aortic valve stenosis
* Kyphoscoliosis
* certain neurological disorders

Exclusion Criteria:

* Patient's refusal to participate in the study
* Psychiatric disorder (impossibility to collect the informed consent)
* Patient under juridical protection
* On going an other study
* Pregnancy, breastfeeding
* Non balanced epilepsy
* 3 grade auriculo-ventricular heart block without pacing
* Severe hepatocellular insufficiency
* Anti arrhythmic treatment : class III of the Vaughan William's classification
* Skin infection of the puncture point
* Allergy to aminoamides local anaesthetic
* Surgical difficulties to insert paravertebral catheter

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2012-10-14 (Actual); Primary Completion 2012-10-14 (Actual); Study Completion 2018-10-11 (Actual)

PRIMARY OUTCOMES:
Total intravenous morphine consumption (mg) | the first 48 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Helms, MD, Principal Investigator
Locations (1):
- Hôpital Civil - NHC Département d'Anesthésiologie, Strasbourg, Alsace, France

REFERENCES:
- [Result] Helms O, Mariano J, Hentz JG, Santelmo N, Falcoz PE, Massard G, Steib A. Intra-operative paravertebral block for postoperative analgesia in thoracotomy patients: a randomized, double-blind, placebo-controlled study. Eur J Cardiothorac Surg. 2011 Oct;40(4):902-6. doi: 10.1016/j.ejcts.2011.01.067. Epub 2011 Mar 5. PMID 21377888